CLINICAL TRIAL: NCT01060215
Title: Clinical Trial for the Effects of Joint Effusion on Proprioception
Brief Title: The Effects of Joint Effusion on Proprioception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: JongIn Lee/Department of Rehabilitation Medicine,, Seoul St. Mary's Hospital, College of Medicine, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 52008B000100044
Record Dates: First submitted 2010-01-28; First posted 2010-02-02 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-01

CONDITIONS: Osteoarthritis
Keywords: effusion; osteoarthritis; knee
MeSH Terms: conditions — Osteoarthritis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Infusion (Active Comparator): 20cc saline infusion into the knee joint
  Interventions: Procedure: Normal saline
- No infusion (No Intervention)
  Interventions: Procedure: Normal saline

INTERVENTIONS:
Procedure: Normal saline — 20 cc normal saline injection into the knee joint

SUMMARY:
The purpose of this study is to assess the effects of joint effusion on proprioceptive status in patients with knee osteoarthritis (OA).

DETAILED DESCRIPTION:
Proprioception is a sensory modality that provides feedback on the internal status of the body and enables us to perceive joint position and motion.

Osteoarthritis (OA), also called degenerative joint disease, is a major musculoskeletal condition characterized by loss of articular cartilage that leads to pain and loss of function. The most commonly affected joint is the knee, and OA may result in changes that affect not only intracapsular tissues, but also periarticular tissues, such as ligaments, capsules, tendons, and muscles. Many studies have examined the proprioceptive status of knee OA, and subjects with knee OA are known to have impaired proprioception compared with age-matched controls.

Joint effusion is a common symptom associated with chronic degenerative joint condition, but the effects of effusion on knee joint proprioception have not been investigated in detail.

A volume of 20 mL of normal saline was injected into the knee joint cavity of subjects in the experimental group under ultrasonographic guidance. Proprioceptive acuity was assessed by active repositioning of the lower limb using an electrogoniometer to measure knee joint position sense (JPS) under both non-weight-bearing and weight-bearing conditions twice, with a 20-min rest interval.

ELIGIBILITY:
Inclusion Criteria:

Or at least two of criteria 2-6 established by the American College of Rheumatology (ACR):

1. Kellgren and Lawrence (K/L) grade ≥II
2. morning stiffness <30 min in duration
3. crepitus on movement of the knee joint
4. bony tenderness at the knee joint margins
5. palpable or visible bony enlargement
6. no palpable warmth.

Exclusion Criteria:

1. the presence of knee joint effusion determined by ultrasonography
2. a history of knee injury or surgery
3. a history of knee injection within 3 months
4. a history of inflammatory arthritis
5. taking anticoagulants
6. balance or gait disturbance
7. diabetes mellitus.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-05; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Proprioceptive acuity in Knee Joint. Proprioceptive acuity (difference between the knee angles at the target and reproduced positions) was assessed by active repositioning of the lower limb after injection or no injection. | within one hour after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jongin Lee, M.D, Study Chair — Department of Rehabilitation Medicine, Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Cho YR, Hong BY, Lim SH, Kim HW, Ko YJ, Im SA, Lee JI. Effects of joint effusion on proprioception in patients with knee osteoarthritis: a single-blind, randomized controlled clinical trial. Osteoarthritis Cartilage. 2011 Jan;19(1):22-8. doi: 10.1016/j.joca.2010.10.013. Epub 2010 Oct 27. PMID 21034839